CLINICAL TRIAL: NCT04658251
Title: Functional Study of Intronic Variants in Inherited Cone Disorders
Brief Title: Study of New Mutations in Cone Disorders
Acronym: INTROCONE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_66; 2020-A02559-30 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Retinal Dystrophy, Cone-Rod; Cone Dystrophy; Cone Rod Dystrophy; Macular Degeneration
Keywords: intronic variant; splicing; functional test; cone disorders; retinal dystrophy; RNA; minigene splice assay; cells
MeSH Terms: conditions — Cone-Rod Dystrophies; Cone Dystrophy; Macular Degeneration; Retinal Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples:
  * Paxgen tubes (2 x 5ml) and heparin tubes (2 x 7ml) will be collected (maximum 32 ml) for RNA extraction if the candidate gene is expressed in the leucocytes
  * Potentially 2 Vacutainer CPT tubes for IPSC generation
  Biopsy:
  Potentially a skin biopsy (3 mm diameter) will be carried out if the gene is not expressed in leucocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an intronic variant unknown in a gene implicated in cone disorders.
  Interventions: Genetic: Blood and/or skin biopsy

INTERVENTIONS:
Genetic: Blood and/or skin biopsy — Blood and/or skin biopsy will be withdrawn, for RNA extraction in order to test the effect of the variant on splicing.

SUMMARY:
High throughput sequencing gives the opportunity to improve the genetic diagnosis for patients suffering from retinal dystrophies and specially from cone disorders. However, a large number of mutations are identified, mostly in introns of the genes, and in silico analysis are not sufficient to assign the pathogenicity of these mutations, without which the diagnosis confirmation cannot be done. For that purpose, a functional analysis of intronic variants of unknown significance detected in patients, with minigene splice assays in parallel with the analysis of the effect of the variant on splicing directly in the cells of the patient, by analyzing the RNA from leucocytes, fibroblasts, lymphoblastoïd cells or precursor of photoreceptor cells, which is the only proof of pathogenicity for variants

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cone disorder
* identification of a variant of unknown significance
* possibility of samplings
* informed consent

Exclusion Criteria:

* no variant of unknown significance identified
* no informed consent

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients carrying an intronic variant of unknown significance (or carrying an exonic variant with a predicted effect on splicing) in a gene implicated (or potentially implicated) in cone disorders, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Effect of the intronic variant on RNA splicing observed in cellulo and/or on patient cells, | at 2 years
  Analysis of RNA transcripts of the gene carrying a variant of unknown significance.

SECONDARY OUTCOMES:
Effect of the intronic variant on RNA by Minigene splice assay in transient cell cultures | at 2 years
Effect of the intronic variant on RNA by analysis of patient RNA transcripts | at 2 years
Effect of the intronic variant on RNA by analysis of transcripts from fibroblasts | at 2 years
Effect of the intronic variant on RNA by analysis of transcripts from lymphoblastoid lines | at 2 years
Effect of the intronic variant on RNA by analysis of transcripts from IPSCs (induced pluripotent stem cells) | at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Claire-Marie DHAENENS, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU lille, Lille, France